CLINICAL TRIAL: NCT02431585
Title: Prevalence of Gluten Sensitivity in Irritable Bowel Syndrome: The First Study in Paediatrics. (GS-IBS)
Brief Title: Prevalence of Gluten Sensitivity in Irritable Bowel Syndrome: The First Study in Paediatrics.
Acronym: GS-IBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Ruggiero Francavilla, MD, PHD, University of Bari
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: GS-IBS
Record Dates: First submitted 2014-10-17; First posted 2015-05-01 (Estimated); Last update posted 2015-05-01 (Estimated); Status verified 2015-04

CONDITIONS: Irritable Bowel Syndrome; Gluten Sensitivity
Keywords: abdominal pain; gluten free diet; functional gastrointestinal disorders
MeSH Terms: conditions — Irritable Bowel Syndrome; Celiac Disease; Abdominal Pain; Gastrointestinal Diseases | interventions — Glutens

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rechallenge (Other): Double blind placebo controlled cross over
  Interventions: Dietary Supplement: gluten; Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: gluten
Dietary Supplement: placebo

SUMMARY:
Recently a new clinical entity, gluten sensitivity (GS), a form of gluten intolerance in which neither allergic nor autoimmune mechanisms can be identified, has been added to the spectrum of gluten-related disorders. This condition is characterized by gastrointestinal and extra-intestinal symptoms including abdominal pain (68%); eczema or rash (40%); headache (35%); diarrhoea (33%) and fatigue (33%). The small intestine of GS patient is usually normal. The prevalence of GS is not yet established although it is estimated that up to 6% of the general population might be affected. GS has been described only in adults and no data are available for the paediatric population.The main problem with this new condition is that, at present, there are no speciﬁc biomarkers to conﬁrm GS diagnosis. In the absence of a serological or histological marker, the diagnosis remains clinical. In order to avoid placebo effect of the dietary treatment, presently GS diagnosis needs to performed with double-blind randomized placebo-controlled challenge provided that both wheat allergy and CD have previously been excluded.

The primary aim of the study is to evaluate the prevalence of GS in IBS paediatric patients.

The secondary aims are: 1) to describe clinical, serologic, genetic and histological profile of GS patient and 2) to study the role of gluten or other possible wheat components in the onset of GS.

Study design Randomized double blind placebo controlled cross over re-challenge trial. Patient consecutively diagnosed as having IBS (Rome III criteria) in whom the diagnosis of coeliac disease and wheat allergy has been excluded, will be considered eligible for the study.

Diagnosis of coeliac disease and wheat allergy will be excluded by the negativity of TTG-IgA and/or EMA and of Skin Prick Test, RAST immuno-CAP and Atopy patch test respectively.

Patients will entered a three-phase study with a running in phase (phase I: weeks 1-2), diagnostic elimination diet phase (phase II: week 3-4) and re-challenge phase (phase III: week 5-12)

DETAILED DESCRIPTION:
Randomized double blind placebo controlled cross over re-challenge trial. Patient consecutively diagnosed as having IBS (Rome III criteria) in whom the diagnosis of coeliac disease and wheat allergy has been excluded, will be considered eligible for the study.

Diagnosis of coeliac disease and wheat allergy will be excluded by the negativity of TTG-IgA and/or EMA and of Skin Prick Test, RAST immuno-CAP and Atopy patch test respectively.

Patients will entered a three-phase study with a running in phase (phase I: weeks 1-2), diagnostic elimination diet phase (phase II: week 3-4) and re-challenge phase (phase III: week 5-12).

The following procedure will be performed at different times (Table 1):

1. Entry (Time 0): Blood test, HLA on blood spot, collection of urine and stools;
2. Running-in (phase I: week 1-2): Visual Analogue Scale (VAS) and (IBS-SS); STAIC test; Bristol stool chart (mBSFC), extra-intestinal symptoms questionnaire.

   At the end of week 2 patients still complaining IBS symptoms (IBS-SS>75) will proceed in the trial and undergo endoscopy plus biopsies on voluntary basis.
3. Diagnostic gluten elimination diet phase (phase II: week 3-4): Visual Analogue Scale (VAS) and (IBS-SS); STAIC test; Bristol stool chart (mBSF-C), extra-intestinal symptoms questionnaire. Collection of urine and stools (end of week 4).

   At the end of week 4 only patients with a significant reduction of IBS symptoms or VAS (greater than 30%) will proceed in the re-challenge phase.

   The challenge phase will be subdivided in Two phases: one double blind phase (product A and B) plus a single blind phase (product C).
4. Product A (week 5-6): Visual Analogue Scale (VAS) and (IBS-SS), STAIC test; Bristol stool chart (mBSF-C), extra-intestinal symptoms questionnaire, collection of urine and stools (end of week 6);
5. Product B (week 8-9): Visual Analogue Scale (VAS) and (IBS-SS), STAIC test; Bristol stool chart (mBSF-C), extra-intestinal symptoms questionnaire, collection of urine and stools (end of week 9)
6. Product C (week 11-12): Visual Analogue Scale (VAS) and (IBS-SS), STAIC test; Bristol stool chart (mBSF-C), extra-intestinal symptoms questionnaire, collection of urine and stools (end of week 12)

Challenge procedure

Double Blind phase (Product A and B):

Children will be asked to keep following the strict gluten free diet and to take a sachet daily for a period of two weeks each interspersed by a washout phase of one week. Sachet will contain either pure gluten (10 grams daily) or gluten free flour (10 grams daily - SHAR). Sachets containing placebo will have the same shape, dimension, indication and appearance as those containing the gluten and will be provided by a bagging factory, which will ensure that the study will be blinded for investigators and patients. Sachets will be named A or B.

Single Blind Challenge (Product C):

To assess whether other components of wheat other gluten are involved in the onset of GS, children will be asked to take for a period of two weeks, while on gluten free diet, a muffin made of wheat flour in a single blind fashion.

ELIGIBILITY:
Inclusion Criteria:

* Age 4-18 years;
* IBS diagnosis according to Roma III criteria;
* Written informed consent.

Exclusion Criteria:

* Coeliac disease;
* Wheat allergy;
* Others food allergy;
* Type 1 Diabetes;
* Others Chronic and or Malignant diseases;
* H. Pylori infection.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The standardized questionnaire (IBS-SS) | 12 weeks
  The severity of IBS symptoms
Visual Analog Scale (VAS) | 12 weeks
Quality of life Questionnaire | 12 weeks
The Faces Pain Scale (FPS) | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Department "B Trambusti" Ospedale Giovanni XXIII Via Amendola 270, Bari, Ba, Italy

REFERENCES:
- [Background] Biesiekierski JR, Peters SL, Newnham ED, Rosella O, Muir JG, Gibson PR. No effects of gluten in patients with self-reported non-celiac gluten sensitivity after dietary reduction of fermentable, poorly absorbed, short-chain carbohydrates. Gastroenterology. 2013 Aug;145(2):320-8.e1-3. doi: 10.1053/j.gastro.2013.04.051. Epub 2013 May 4. PMID 23648697
- [Background] Biesiekierski JR, Newnham ED, Irving PM, Barrett JS, Haines M, Doecke JD, Shepherd SJ, Muir JG, Gibson PR. Gluten causes gastrointestinal symptoms in subjects without celiac disease: a double-blind randomized placebo-controlled trial. Am J Gastroenterol. 2011 Mar;106(3):508-14; quiz 515. doi: 10.1038/ajg.2010.487. Epub 2011 Jan 11. PMID 21224837
- [Background] Volta U, Bardella MT, Calabro A, Troncone R, Corazza GR; Study Group for Non-Celiac Gluten Sensitivity. An Italian prospective multicenter survey on patients suspected of having non-celiac gluten sensitivity. BMC Med. 2014 May 23;12:85. doi: 10.1186/1741-7015-12-85. PMID 24885375
- [Background] Catassi C, Bai JC, Bonaz B, Bouma G, Calabro A, Carroccio A, Castillejo G, Ciacci C, Cristofori F, Dolinsek J, Francavilla R, Elli L, Green P, Holtmeier W, Koehler P, Koletzko S, Meinhold C, Sanders D, Schumann M, Schuppan D, Ullrich R, Vecsei A, Volta U, Zevallos V, Sapone A, Fasano A. Non-Celiac Gluten sensitivity: the new frontier of gluten related disorders. Nutrients. 2013 Sep 26;5(10):3839-53. doi: 10.3390/nu5103839. PMID 24077239
- [Background] Carroccio A, Mansueto P, Iacono G, Soresi M, D'Alcamo A, Cavataio F, Brusca I, Florena AM, Ambrosiano G, Seidita A, Pirrone G, Rini GB. Non-celiac wheat sensitivity diagnosed by double-blind placebo-controlled challenge: exploring a new clinical entity. Am J Gastroenterol. 2012 Dec;107(12):1898-906; quiz 1907. doi: 10.1038/ajg.2012.236. Epub 2012 Jul 24. PMID 22825366
- [Derived] Francavilla R, Cristofori F, Verzillo L, Gentile A, Castellaneta S, Polloni C, Giorgio V, Verduci E, D'Angelo E, Dellatte S, Indrio F. Randomized Double-Blind Placebo-Controlled Crossover Trial for the Diagnosis of Non-Celiac Gluten Sensitivity in Children. Am J Gastroenterol. 2018 Mar;113(3):421-430. doi: 10.1038/ajg.2017.483. Epub 2018 Jan 30. PMID 29380821